CLINICAL TRIAL: NCT04161209
Title: The Effect of Acute Citalopram on Response to Acute Stress Induction
Brief Title: Citalopram and Stress Reactivity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Oxford (Other)
Collaborators: University of Bath (Other)
Responsible Party: Principal Investigator, drsusannahmurphy, Senior Research Fellow, University of Oxford
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: OCST_Citalopram
Record Dates: First submitted 2019-11-08; First posted 2019-11-13 (Actual); Last update posted 2019-11-15 (Actual); Status verified 2019-11

CONDITIONS: Depression; Depressive Disorder; Mental Disorder; Antidepressive Agents; Cognition; Stress
Keywords: Citalopram; Stress induction paradigm; Healthy volunteers
MeSH Terms: conditions — Depression; Depressive Disorder; Mental Disorders | interventions — Citalopram

STUDY DESIGN:
Intervention Model Description: Following the screening, eligible participants will be randomised to receive either a single 20mg oral dose of citalopram or a matched lactose placebo tablet using an online randomisation tool. Note that the study is not assessing the safety or efficacy of citalopram, rather it is using citalopram to understand the role of serotonin in stress reactivity.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drug: Citalopram (Experimental): 20mg oral dose of citalopram (tablet encapsulated in opaque capsule)
  Interventions: Drug: Citalopram
- Placebo (Placebo Comparator): Lactose placebo (tablet encapsulated in opaque capsule)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Citalopram — Single dose administration of citalopram (20mg)
  Arms: Drug: Citalopram
Other: Placebo — Lactose placebo tablet
  Arms: Placebo

SUMMARY:
This study is investigating whether acute administration of citalopram is associated with a decrease in stress reactivity in healthy volunteers, compared to placebo administration. Using a parallel-group double-blind design, participants will be randomised to receive either an acute dose of citalopram or placebo. All participants will have come in for a screening visit. On the day of the research visit (following drug administration) participants will have completed a number of widely used computer-based cognitive tasks measuring emotional processing biases. They will then complete the Oxford Cognition Stress Task, a web-based acute stress induction paradigm, which is designed to induce mild transient increases in stress and arousal. Identifying early changes in stress reactivity following antidepressant treatment will increase the investigator's knowledge of how antidepressants operate, and provide putative targets to identify early response to antidepressants.

DETAILED DESCRIPTION:
In the Oxford Cognition Stress Task (OCST), participants are presented with a series of mental arithmetic, verbal (anagrams) and visuospatial (visual search) challenges on a computer screen. There is a time limit for completing each challenge, which is displayed on the screen as a time bar. To induce a high failure rate, the timing and difficulty of the challenges is automatically varied to ensure participants are correctly complete only 20-40% of the challenges within the time, and some of the verbal challenges (anagrams) are impossible to solve. Participants are given feedback on their performance on the screen which indicates that they are performing badly. Heart rate will be measured continuously during the OCST, and during pre- and post- task periods. Baseline and post-OCST measures of blood pressure and samples of saliva (for cortisol analysis) will be taken. Participants will also complete Visual Analogue Scales pre- and post-OCST to give a subjective measure of stress and mood. Participants will not be told the extent to which becoming stressed (and finding the task difficult) is intended. At the end of the test session, participants will be fully debriefed as to the nature of the OCST.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female
* Aged 18 -45 years
* Fluent in written and spoken English at a sufficient level to understand and complete the tasks
* Body Mass Index (BMI) 18-30
* Participant is willing and able to give informed consent for participation in the study
* Not currently taking any regular medications (expect the contraceptive pill)

Exclusion Criteria:

* Any past or current Axis 1 DSM-V psychiatric disorder
* Current use of psychoactive medication (except the contraceptive pill, the Depo-Provera injection or the progesterone implant) or medication which may affect the stress response (e.g. corticosteroids, beta-blockers)
* Current or past history of drug or alcohol dependency
* History of current significant neurological condition (e.g. epilepsy) or heart disease/hypertension
* Known hypersensitivity to the study drug
* Currently pregnant or breast feeding
* Previous participation in a study that uses the same or similar computer tasks as those used in the present study
* Previous participation in a study that involves the use of a medication within the last three months
* Significant medical condition
* Smokers consuming > 5 cigarettes per day
* Individuals consuming > 6 caffeinated drinks per day
* Lactose Intolerance (due to the study involving administration of a lactose placebo tablet)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-10-11 (Actual); Primary Completion 2020-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Heart rate (beats per minute) | Day 1: 4.5-5.5 hours post drug administration
  Difference in heart rate during the Oxford Cognition Stress Task relative to pre-task baseline period between citalopram and placebo groups

SECONDARY OUTCOMES:
Heart rate variability (Root Mean Square Of Successive Differences: RMSSD) | Day 1: 4.5-5.5 hours post drug administration
  Difference in RMSSD during the Oxford Cognition Stress Task relative to pre-task baseline period between citalopram and placebo groups
Salivary cortisol | Day 1: 4.5-5.5 hours post drug administration
  Difference in salivary cortisol following the Oxford Cognition Stress Task relative to pre-task baseline between citalopram and placebo groups; difference in area under the curve for all study timepoints between citalopram and placebo groups
Blood pressure | Day 1: 4.5-5.5 hours post drug administration
  Difference in systolic and diastolic blood pressure following the Oxford Cognition Stress Task relative to pre-task baseline between citalopram and placebo groups
Subjective measures of stress and arousal | Day 1: 4.5-5.5 hours post drug administration
  Difference in state anxiety, positive and negative affect, and Visual Analogue Scale (VAS) ratings of stress (from 0 to 100, where 0 indicates 'Not at all' and 100 indicates 'Extremely') following the Oxford Cognition Stress Task relative to pre-task baseline between citalopram and placebo groups

CONTACTS AND LOCATIONS:
Overall Officials: Susannah Murphy, DPhil, Principal Investigator — University of Oxford
Locations (1):
- University of Oxford, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
An anonymised dataset will be published as open access data on a secure repository (Open Science Framework https://osf/io/).
Supporting Information: Study Protocol, ICF
Time Frame: Following full anonymisation of study data and publication of findings. Data will be stored indefinitely.

REFERENCES:
- See also: PERL Oxford webpage — http://www.psych.ox.ac.uk/research/psychopharmacology-and-emotion-research-laboratory